CLINICAL TRIAL: NCT00932750
Title: THE EFFECTS OF COFFEE MANNOOLIGOSACCHARIDES ON INDICES OF BODY WEIGHT, BODY COMPOSITION, AND SATIETY IN HUMANS
Brief Title: Study of Coffee Mannooligosaccharides for Weight Management
Acronym: MOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Marie-Pierre St-Onge, Ph.D Research Associate, St. Luke's/Roosevelt Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KF-MOS-01
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: Body composition; Weight loss; Weight management; Beverages; Diet
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOS Weight maintenance (Placebo Comparator)
  Interventions: Dietary Supplement: Coffee mannooligosaccharide
- MOS weight loss (Placebo Comparator)
  Interventions: Dietary Supplement: Coffee mannooligosaccharides

INTERVENTIONS:
Dietary Supplement: Coffee mannooligosaccharide — 2 beverages daily providing either 4 g of coffee mannooligosaccharide or placebo.
  Arms: MOS Weight maintenance
Dietary Supplement: Coffee mannooligosaccharides — Subjects consume 2 beverages daily providing 4 g of coffee mannooligosaccharides or placebo
  Arms: MOS weight loss

SUMMARY:
The goal of this study is to establish the role of coffee mannooligosaccharides (MOS), provided in a beverage format, on body weight regulation. Overweight and obese men and women will be randomized to one of 2 groups: placebo or MOS beverage. They will be required to consume 2 beverages/day for the duration of the 2 phases of the study. The MOS beverage will provide 2 g of MOS (total of 4 g/d). This dose level has been found to be well tolerated and safe. In the first phase, subjects will be counseled once monthly on a nutrition-related topic on an individual basis. They will be asked to maintain their regular eating and exercise habits for the duration of the 12 week period. An 8-week washout period will follow during which time they will not be required to consume the beverages. The second phase of the study will be a weight loss phase. For this phase, subjects will be re-randomized and may consume the alternate or the same beverage as the first phase, depending on the outcome of randomization. During this phase, they will undergo group counseling on a weekly basis. Counseling sessions will focus on weight loss and ways to achieve moderate weight loss of approximately 1-2 lbs/week. Measurements will be taken at the beginning and end of each phase. This study will allow us to determine whether MOS helps maintain body weight and prevent weight gain (first phase) and whether it helps to stimulate weight loss (second phase). The results will allow us to find ways in which overweight and obese individuals can incorporate beverages in their diets that will help promote weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 27-33 kg/m2
* Stable body weight

Exclusion Criteria:

* Body width > 46 cm
* Medications known to affect body weight, lipids, blood pressure
* Pregnant or lactating women
* Less than 1 y post-partum

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Body Composition by Magnetic Resonance Imaging | Baseline and Endpoint
Blood pressure | Weekly
Body weight | Weekly
Waist circumference | Weekly

SECONDARY OUTCOMES:
Appetite/Satiety | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Ph.D, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's/Roosevelt Hospital, New York, New York, United States